CLINICAL TRIAL: NCT01241032
Title: A Randomized, Open, Crossover Clinical Study to Investigate the Effects of Alcohol on the Pharmacokinetics of Udenafil Tablet in Healthy Male Volunteers
Brief Title: Phase I Study to Investigate the Alcohol Interaction of DA8159
Acronym: DA8159_DIA_I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Clinical Development Team1, Dong-A Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-0086
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers; Erectile Dysfunction
Keywords: DA-8159; Udenafil; Alcohol
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Udenafil (Experimental): Udenafil 200mg
  Interventions: Drug: Udenafil
- Udenafil + Alcohol (Active Comparator): Udenafil 200mg + Alcohol
  Interventions: Drug: Udenafil; Dietary Supplement: Alcohol

INTERVENTIONS:
Drug: Udenafil — 200mg Single Oral Dose of
Dietary Supplement: Alcohol — Alcohol 39g / 240ml
  Arms: Udenafil + Alcohol

SUMMARY:
This study is designed to to investigate the effects of alcohol on the pharmacokinetics of Udenafil tablet in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 19 to 55 years at screening.
* Subjects with body weight ≥ 55 kg and within ±20% of the ideal body weight : Ideal body weight = (height [cm] - 100)x0.9.
* Subjects who have received and understood completely the information regarding the current study and given written informed consents to voluntarily participate in the study and followed all instructions specified in the protocol.

Exclusion Criteria:

* Subjects with the test results of QTc > 430 ms or non-sinus cardiac rhythm by ECG analysis.
* Subjects with hypotension or hypertension.
* Subjects who have drunken habitually (exceeding 21 units/week, 1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the study period from 2 days prior to the first administration of investigational product and during this study.
* Subjects deemed ineligible by investigator based on other reasons, including abnormal laboratory values or diseases.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Cmax) | 48 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: Clinical Research Center, Asan Medical Center — http://crc.amc.seoul.kr